CLINICAL TRIAL: NCT01890096
Title: A Randomized Phase II Trial of High Dose-Rate Brachytherapy as Monotherapy in Low and Intermediate Risk Prostate Cancer
Brief Title: A Phase II Trial of High Dose-Rate Brachytherapy as Monotherapy in Low and Intermediate Risk Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gerard Morton, Dr. Gerard Morton, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMOR_HDR Monotherapy RCT
Record Dates: First submitted 2013-06-26; First posted 2013-07-01 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Carcinoma of the Prostate
Keywords: HDR; monotherapy; low; intermediate; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HDR 2 fractions (Experimental): HDR brachytherapy of 27 Gy delivered in 2 fractions one week apart
  Interventions: Radiation: HDR 2 Fraction
- HDR 1 fraction (Experimental): HDR brachytherapy of 19 Gy delivered in a single fraction
  Interventions: Radiation: HDR 1 Fraction

INTERVENTIONS:
Radiation: HDR 2 Fraction — High dose-rate brachytherapy using real-time intra-operative transrectal ultrasound guidance. Patients will receive 27 Gy as a minimal Clinical Target Volume (CTV) dose delivered as two fractions of 13.5 Gy 7-13 days apart. The CTV is the ultrasound defined prostate with a 0-2 mm margin.
  Arms: HDR 2 fractions
Radiation: HDR 1 Fraction — High Dose-Rate Brachytherapy delivered in same manner as Arm 1, but to a prescribed CTV minimal dose of 19 Gy in a single fraction
  Arms: HDR 1 fraction

SUMMARY:
A single high dose rate brachytherapy (HDR) treatment combined with a short course of external beam radiotherapy (EBRT) is a highly effective and well tolerated treatment for men with intermediate risk prostate cancer. High cancer control rates have also been reported with HDR used on its own, without the EBRT. The challenge has been to determine what HDR dose to use with a move towards one or two fractions by several investigators. These schedules are reported to be well tolerated in the short term, but with little long term data. The objective of this study is to investigate HDR monotherapy given as either one fraction of 19 Gy or two fractions of 13.5 Gy in a randomized phase II clinical trial. The primary endpoint is patient reported toxicity and health related quality of life at 1 year, and efficacy data will be also be analyzed. Sample size for the study is 174 patients, which we expect to accrue within 18 months.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of adenocarcinoma of the prostate
* low and intermediate risk disease defined as either Gleason 6 or Gleason 7 and PSA < 20ng/mL. PSA to be drawn within 60 days of registration
* prostate volume < 60 cc as determined by ultrasound, CT or MRI
* willing to give informed consent ot participate in this clinical trial
* able and willing to complete Expanded Prostate Index Composite (EPIC) questionnaire

Exclusion Criteria:

* documented nodal or distant metastases
* previous pelvic radiotherapy
* previous trans-urethral resection of prostate, previous prostatectomy or Highly Focused Ultrasound (HIFU)
* use of androgen deprivation therapy. Use of 5-alpha reductase inhibitors is permitted
* poor baseline urinary function defined as radiotherapy eg. connective tissue disease or inflammatory bowel disease
* significant medical co-morbidity rendering patient unsuitable for general anaesthetic

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-05-01 (Actual); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life (QoL) | 1 year
  To demonstrate that health related QoL at 1 year in the urinary and bowel domains of the Expanded Prostate Index Composite (EPIC) for at least one HDR monotherapy arm is not worse than that following current standard treatment with single fraction HDR combined with supplemental external beam radiotherapy.

SECONDARY OUTCOMES:
GU and GI toxicities | baseline, 6 weeks post treament, 3mths, 6mths, 6 monthly for the first 3 years, annually up to 5 years
  To determine genito-urinary (GU) and gastro-intestinal (GI) toxicities in both study arms according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0
Urinary Symptoms | baseline, 6 weeks post treatment, 3 mths, 6 mths, 6-monthly for the first 3 years, annually until 5 years
  To determine changes in urinary symptoms in both study arms as determined by the International Prostate Symptom Score (IPSS)
Serum PSA changes | baseline, 6 weeks post treatment, 3 mths, 6 mths, 6-monthly up to 3 years, annually until 5 years
  To determine changes in serum prostate-specific antigen (PSA) in both arms
Biochemical failure and disease free survival rates | 5 years
  To determine PSA failure and disease free survival rates in both study arms
Erectile function | 5 year
  To determine changes in erectile function in both study arms assessed using the International Index of Erectile Function (IIEF) scale
Associations between dosimetric parameters and toxicity/EPIC domains | 5 years
  To explore association between dosimetric parameters and toxicity/EPIC domain change

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Morton, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada